CLINICAL TRIAL: NCT06972095
Title: The Performance of the Endurant Endoprosthesis in an Infrarenal Aortic Aneurysm With a Wide or Conical Shaped Infrarenal Neck Anatomy
Brief Title: Results Wide and Conical Neck EVAR Procedures
Acronym: Endurant_WCN
Status: Completed | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-1830
Record Dates: First submitted 2025-04-17; First posted 2025-05-14 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: abdominal aortic aneurysm; EVAR; wide neck; conical neck; hostile neck
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Wide neck group: patients with an abdominal aortic aneurysm and a wide neck (>28 mm diameter)
  Interventions: Procedure: EVAR
- conical neck group: patients with an abdominal aortic aneurysm and a conical neck
  Interventions: Procedure: EVAR
- straight neck group: patients with an abdominal aortic aneurysm without a wide or conical neck
  Interventions: Procedure: EVAR

INTERVENTIONS:
Procedure: EVAR — endovascular repair of the AAA with the endurant stent graft

SUMMARY:
Retrospective single centre observational cohort study of patients who underwent an elective infrarenal abdominal aortic aneurysm repair, from January 2011 to January 2020.

DETAILED DESCRIPTION:
Objective: To evaluate the performance of the Endurant endoprothesis in patients with a wide or conical shaped neck anatomy after elective abdominal aortic aneurysm repair.

Inclusion: Patients who underwent elective infrarenal abdominal aortic aneurysm repair with the Endurant endograft between January 2011 until January 2020 in Rijnstate, Arnhem, the Netherlands.

Primary endpoint: Freedom from reinterventions at one year.

Secondary outcomes:

* Endoleaks
* Aneurysm sac growth
* Aneurysm rupture
* Stent migration
* AAA-related mortality
* All-cause mortality
* Procedural time
* 30-day complications
* Renal dysfunction/renal occlusion
* Proximal fixation failure

ELIGIBILITY:
Inclusion Criteria:

All patients with an elective infrarenal endovascular abdominal aortic aneurysm repair with the Endurant endoprothesis between January 2011 till January 2020 in the Rijnstate hospital, Arnhem, the Netherlands.

Exclusion Criteria:

* emergency/rupture procedures
* objection use of data for research
* other prosthesis used for EVAR

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with an elective infrarenal endovascular abdominal aortic aneurysm repair with the Endurant endoprothesis between January 2011 till January 2020 in the Rijnstate hospital, Arnhem, the Netherlands.
Sampling Method: Non-Probability Sample
Enrollment: 268 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2025-04-17 (Actual)

PRIMARY OUTCOMES:
Freedom from reinterventions at one year | one year
  reintervention-free survival will be evaulated using kaplan meier method

SECONDARY OUTCOMES:
Freedom from reinterventions throughout follow-up (up to ten years) | 10 years
  Reintervention-free survival throughout all available follow-up will be evaluated using kaplan-meier methods
Number of endoleaks | 10 year follow-up
  All endoleaks will be registered throughout follow-up and will be presented by type of endoleak.
the number of patients showing aneurysm sac growth | 10 year follow-up
  Sac growth is defined as growth over 5 mm and will be presented for 1 year follow-up, 5 years follow-up and 10 year follow-up
the number of patients with an aneurysm rupture during follow-up | 10 year follow-up
  all ruptures that occur will be registered including outcome (death or successful repair)
the number of patients showing stent migration | 10 year follow-up
  stent migration will be documented in mm and will be presented for 1 year follow-up, 5 years follow-up and 10 year follow-up
Number of patients with AAA related mortality | 10 year follow-up
  All deaths related to the AAA will be documented
the number of patients showing proximal fixation failure | 10 year follow-up
  proximal fixation failure is defined as yes if type 1 endoleak or stent migration or aneurysm sac growth will occur and will be presented for 1 year follow-up, 5 years follow-up and 10 year follow-up
All-cause mortality | 10 year follow-up
  all deaths will be registered regardless their cause
The number of patients with 30-day complications | 30 days
  All complications during the first 30 days will be registered related to the procedure and will be listed for the different types of complications
The number of patients with renal dysfunction/renal occlusion | 10 year follow-up
  all clinical relevant declines in renal function will be documented, including renal artery stenosis or occlusion

CONTACTS AND LOCATIONS:
Overall Officials: M.M.P.J. Reijnen Vascular Surgeon, Prof. Dr., Principal Investigator — Rijnstate
Locations (1):
- Rijnstate, Arnhem, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
On request we can decide if data can be shared; due to country and hospital policy, data transfer agreements need to be in place